CLINICAL TRIAL: NCT01273766
Title: Impact of Intervention With Deferasirox on the Immune Function of Patients With Hematologic Diseases and Transfusion-Related Iron Overload
Brief Title: Deferasirox in Treating Iron Overload Caused By Blood Transfusions in Patients With Hematologic Malignancies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00015287; NCI-2010-02228 (Other Grant/Funding Number: NCI); CCCWFU 97710 (Other: Wake Forest University Health Sciences)
Record Dates: First submitted 2011-01-07; First posted 2011-01-10 (Estimated); Results first posted 2013-11-27 (Estimated); Last update posted 2018-09-07 (Actual); Status verified 2018-08

CONDITIONS: Acute Undifferentiated Leukemia; Adult Acute Lymphoblastic Leukemia in Remission; Adult Acute Myeloid Leukemia in Remission; Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Del(5q); Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(15;17)(q22;q12); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Adult Grade III Lymphomatoid Granulomatosis; Adult Langerhans Cell Histiocytosis; Adult Nasal Type Extranodal NK/T-cell Lymphoma; Anaplastic Large Cell Lymphoma; Angioimmunoblastic T-cell Lymphoma; Contiguous Stage II Adult Burkitt Lymphoma; Contiguous Stage II Adult Diffuse Large Cell Lymphoma; Contiguous Stage II Adult Diffuse Mixed Cell Lymphoma; Contiguous Stage II Adult Diffuse Small Cleaved Cell Lymphoma; Contiguous Stage II Adult Immunoblastic Large Cell Lymphoma; Contiguous Stage II Adult Lymphoblastic Lymphoma; Contiguous Stage II Grade 1 Follicular Lymphoma; Contiguous Stage II Grade 2 Follicular Lymphoma; Contiguous Stage II Grade 3 Follicular Lymphoma; Contiguous Stage II Mantle Cell Lymphoma; Contiguous Stage II Marginal Zone Lymphoma; Contiguous Stage II Small Lymphocytic Lymphoma; Cutaneous B-cell Non-Hodgkin Lymphoma; de Novo Myelodysplastic Syndromes; Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Hepatosplenic T-cell Lymphoma; Intraocular Lymphoma; Mast Cell Leukemia; Myelodysplastic Syndrome With Isolated Del(5q); Myelodysplastic/Myeloproliferative Neoplasm, Unclassifiable; Myeloid/NK-cell Acute Leukemia; Nodal Marginal Zone B-cell Lymphoma; Noncontiguous Stage II Adult Burkitt Lymphoma; Noncontiguous Stage II Adult Diffuse Large Cell Lymphoma; Noncontiguous Stage II Adult Diffuse Mixed Cell Lymphoma; Noncontiguous Stage II Adult Diffuse Small Cleaved Cell Lymphoma; Noncontiguous Stage II Adult Immunoblastic Large Cell Lymphoma; Noncontiguous Stage II Adult Lymphoblastic Lymphoma; Noncontiguous Stage II Grade 1 Follicular Lymphoma; Noncontiguous Stage II Grade 2 Follicular Lymphoma; Noncontiguous Stage II Grade 3 Follicular Lymphoma; Noncontiguous Stage II Mantle Cell Lymphoma; Noncontiguous Stage II Marginal Zone Lymphoma; Noncontiguous Stage II Small Lymphocytic Lymphoma; Noncutaneous Extranodal Lymphoma; Peripheral T-cell Lymphoma; Previously Treated Myelodysplastic Syndromes; Primary Myelofibrosis; Recurrent Adult Acute Lymphoblastic Leukemia; Recurrent Adult Acute Myeloid Leukemia; Recurrent Adult Burkitt Lymphoma; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Adult Diffuse Mixed Cell Lymphoma; Recurrent Adult Diffuse Small Cleaved Cell Lymphoma; Recurrent Adult Grade III Lymphomatoid Granulomatosis; Recurrent Adult Hodgkin Lymphoma; Recurrent Adult Immunoblastic Large Cell Lymphoma; Recurrent Adult Lymphoblastic Lymphoma; Recurrent Adult T-cell Leukemia/Lymphoma; Recurrent Cutaneous T-cell Non-Hodgkin Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Mycosis Fungoides/Sezary Syndrome; Recurrent Small Lymphocytic Lymphoma; Refractory Anemia; Refractory Multiple Myeloma; Secondary Acute Myeloid Leukemia; Secondary Myelofibrosis; Small Intestine Lymphoma; Splenic Marginal Zone Lymphoma; Stage I Adult Burkitt Lymphoma; Stage I Adult Diffuse Large Cell Lymphoma; Stage I Adult Diffuse Mixed Cell Lymphoma; Stage I Adult Diffuse Small Cleaved Cell Lymphoma; Stage I Adult Hodgkin Lymphoma; Stage I Adult Immunoblastic Large Cell Lymphoma; Stage I Adult Lymphoblastic Lymphoma; Stage I Adult T-cell Leukemia/Lymphoma; Stage I Cutaneous T-cell Non-Hodgkin Lymphoma; Stage I Grade 1 Follicular Lymphoma; Stage I Grade 2 Follicular Lymphoma; Stage I Grade 3 Follicular Lymphoma; Stage I Mantle Cell Lymphoma; Stage I Marginal Zone Lymphoma; Stage I Multiple Myeloma; Stage I Mycosis Fungoides/Sezary Syndrome; Stage I Small Lymphocytic Lymphoma; Stage II Adult Hodgkin Lymphoma; Stage II Adult T-cell Leukemia/Lymphoma; Stage II Cutaneous T-cell Non-Hodgkin Lymphoma; Stage II Multiple Myeloma; Stage II Mycosis Fungoides/Sezary Syndrome; Stage III Adult Burkitt Lymphoma; Stage III Adult Diffuse Large Cell Lymphoma; Stage III Adult Diffuse Mixed Cell Lymphoma; Stage III Adult Diffuse Small Cleaved Cell Lymphoma; Stage III Adult Hodgkin Lymphoma; Stage III Adult Immunoblastic Large Cell Lymphoma; Stage III Adult Lymphoblastic Lymphoma; Stage III Adult T-cell Leukemia/Lymphoma; Stage III Cutaneous T-cell Non-Hodgkin Lymphoma; Stage III Grade 1 Follicular Lymphoma; Stage III Grade 2 Follicular Lymphoma; Stage III Grade 3 Follicular Lymphoma; Stage III Mantle Cell Lymphoma; Stage III Marginal Zone Lymphoma; Stage III Multiple Myeloma; Stage III Mycosis Fungoides/Sezary Syndrome; Stage III Small Lymphocytic Lymphoma; Stage IV Adult Burkitt Lymphoma; Stage IV Adult Diffuse Large Cell Lymphoma; Stage IV Adult Diffuse Mixed Cell Lymphoma; Stage IV Adult Diffuse Small Cleaved Cell Lymphoma; Stage IV Adult Hodgkin Lymphoma; Stage IV Adult Immunoblastic Large Cell Lymphoma; Stage IV Adult Lymphoblastic Lymphoma; Stage IV Adult T-cell Leukemia/Lymphoma; Stage IV Cutaneous T-cell Non-Hodgkin Lymphoma; Stage IV Grade 1 Follicular Lymphoma; Stage IV Grade 2 Follicular Lymphoma; Stage IV Grade 3 Follicular Lymphoma; Stage IV Mantle Cell Lymphoma; Stage IV Marginal Zone Lymphoma; Stage IV Mycosis Fungoides/Sezary Syndrome; Stage IV Small Lymphocytic Lymphoma; Testicular Lymphoma; Untreated Adult Acute Lymphoblastic Leukemia; Untreated Adult Acute Myeloid Leukemia; Waldenstrom Macroglobulinemia
MeSH Terms: conditions — Leukemia, Biphenotypic, Acute; Congenital Abnormalities; Histiocytosis, Langerhans-Cell; Lymphoma, Extranodal NK-T-Cell; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Intraocular Lymphoma; Leukemia, Mast-Cell; Chromosome 5q Deletion Syndrome; Myeloproliferative Disorders; Lymphoma, B-Cell, Marginal Zone; Lymphoma, T-Cell, Peripheral; Primary Myelofibrosis; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Mycosis Fungoides; Sezary Syndrome; Leukemia, Lymphocytic, Chronic, B-Cell; Anemia, Refractory; Multiple Myeloma; Waldenstrom Macroglobulinemia | interventions — Deferasirox; Enzyme-Linked Immunosorbent Assay

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm I (Experimental): Patients receive oral deferasirox once daily for up to 6 months or until blood counts recover in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: deferasirox; Other: laboratory biomarker analysis; Other: enzyme-linked immunosorbent assay
- control arm (No Intervention): blood tested on healthy patients
- correlative (No Intervention): treated off study with or without oral deferasirox (patient choice) but lab draws to gather lab analysis

INTERVENTIONS:
Drug: deferasirox — Given orally
  Other Names: Exjade; ICL670
  Arms: Arm I
Other: laboratory biomarker analysis — Correlative studies
  Arms: Arm I
Other: enzyme-linked immunosorbent assay — Correlative studies
  Other Names: ELISA
  Arms: Arm I

SUMMARY:
RATIONALE: Deferasirox may remove excess iron from the body caused by blood transfusions.

PURPOSE: This clinical trial studies deferasirox in treating iron overload caused by blood transfusions in patients with hematologic malignancies.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES: I. To determine the effects of the iron-chelating agent deferasirox on changes in: neutrophil function; macrophage function; lymphocyte function.

SECONDARY OBJECTIVES: I. To determine the effect of chelation on the incidence of bacterial, viral and fungal infections documented by clinical, microbiologically-proven versus radiologically-proven criteria. II. To determine the effect of iron chelation on mortality and morbidity with incidence of the following parameters: Need for hospitalization; Duration of hospitalization; Need for ventilatory support; Need for exchange transfusion/apheresis; Need for treatment with antifungals or antibiotics for documented infections.

OUTLINE: Patients receive oral deferasirox once daily for up to 6 months or until blood counts recover in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a pathology confirmed diagnosis of one of the following: myelodysplastic syndrome (MDS); acute leukemia; multiple myeloma; myelofibrosis; lymphoma; chronic anemia; sickle cell anemia
* Iron score >= 2
* Absolute Neutrophil Count (ANC) >= 1,000
* Platelets >= 50,000
* Albumin >= 2 g/dL
* Alkaline phosphatase =< 5X Upper Limit of Normal (ULN)
* Total bilirubin =< 1.5
* Creatinine =< 2X age-appropriate Upper Limit of Normal (ULN) OR creatinine clearance >= 40 ml/min
* Serum Glutamic Oxaloacetic Transaminase (SGOT) [AST] and Serum Glutamic Pyruvic Transaminase (SGPT) [ALT] =< 5X Upper Limit of Normal (ULN)
* Eastern Cooperative Oncology Group(ECOG) performance status of 0 or 1
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients with active disease undergoing chemotherapy treatment
* Patient who have been treated with rituximab or immunomodulating drugs =< 1 month prior to enrollment
* HIV-positive patients
* Hepatitis-C positive patients
* Women who are pregnant or breastfeeding
* Patients on hemodialysis/patients with renal failure
* Patients with sepsis or acute illness
* Known hypersensitivity to deferasirox
* Patients with moderate or severe hearing loss as defined by audiogram

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2011-01; Primary Completion 2012-03 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Ann Knovich, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Comprehensive Cancer Center of Wake Forest University, Winston-Salem, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I: Patients receive oral deferasirox once daily for up to 6 months or until blood counts recover in the absence of disease progression or unacceptable toxicity.
  deferasirox : Given orally
  laboratory biomarker analysis : Correlative studies
  enzyme-linked immunosorbent assay : Correlative studies
Period: Overall Study
Arm/Group | Arm I | Control Arm | Correlative
Started | 4 | 7 | 5
Completed | 4 | 7 | 5
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I | Control Arm | Correlative | Total
Number analyzed (Participants) | 4 | 7 | 5 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 7 | 4 | 14
  >=65 years | 1 | 0 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.1 (12.9) | 40.1 (7.0) | 55.0 (17.6) | 48.0 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 6 | 1 | 9
  Male | 2 | 1 | 4 | 7
Region of Enrollment [Number; unit: participants]
  United States | 4 | 7 | 5 | 16

OUTCOME MEASURES:

1. Primary Outcome: Changes in Mean Neutrophil Values (as Measured by Lab) for Arm 1 (Other Arms Were Used for Calibration Only)
Description: Changes in Neutrophils between baseline and mean neutrophils values during treatment (measured after each dose)
Time Frame: Baseline, up to 6 months
Measure: Mean (Standard Deviation); unit: 10^9 Neutrophils per Liter
Arm/Group | Arm I
Number analyzed (Participants) | 4
10^9 Neutrophils per Liter | 7.8 (138.4)

2. Secondary Outcome: Need for Hospitalization, Ventilator Support, Exchange Transfusion/Apheresis or Treatment With Antifungals or Antibiotics
Description: Records will be assessed at baseline and prospectively while on study.
Time Frame: Baseline, up to 6 months
Population: Number analyzed in rows differs from overall because data was not collected on all participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I | Correlative
Number analyzed (Participants) | 4 | 5
Participants
  Baseline : Hospitalization: number analyzed (Participants) | 2 | 5
  Baseline : Hospitalization | 2 | 5
  Baseline : Ventilator: number analyzed (Participants) | 2 | 5
  Baseline : Ventilator | 0 | 1
  Baseline : Transfusion: number analyzed (Participants) | 2 | 5
  Baseline : Transfusion | 0 | 0
  Baseline : Antibiotics: number analyzed (Participants) | 2 | 5
  Baseline : Antibiotics | 0 | 5
  1 Month : Hospitalization: number analyzed (Participants) | 3 | 3
  1 Month : Hospitalization | 1 | 1
  1 Month : Ventilator: number analyzed (Participants) | 3 | 3
  1 Month : Ventilator | 0 | 0
  1 Month : Transfusion: number analyzed (Participants) | 3 | 3
  1 Month : Transfusion | 0 | 1
  1 Month : Antibiotics: number analyzed (Participants) | 3 | 3
  1 Month : Antibiotics | 1 | 1
  2 Month : Hospitalization: number analyzed (Participants) | 4 | 3
  2 Month : Hospitalization | 0 | 1
  2 Month : Ventilator: number analyzed (Participants) | 4 | 3
  2 Month : Ventilator | 0 | 0
  2 Month : Transfusion: number analyzed (Participants) | 4 | 3
  2 Month : Transfusion | 0 | 1
  2 Month : Antibiotics: number analyzed (Participants) | 4 | 3
  2 Month : Antibiotics | 0 | 1
  3 Month : Hospitalization: number analyzed (Participants) | 4 | 4
  3 Month : Hospitalization | 0 | 1
  3 Month : Ventilator: number analyzed (Participants) | 4 | 4
  3 Month : Ventilator | 0 | 0
  3 Month : Transfusion: number analyzed (Participants) | 4 | 4
  3 Month : Transfusion | 0 | 1
  3 Month : Antibiotics: number analyzed (Participants) | 4 | 4
  3 Month : Antibiotics | 0 | 0
  4 Month : Hospitalization: number analyzed (Participants) | 4 | 3
  4 Month : Hospitalization | 0 | 1
  4 Month : Ventilator: number analyzed (Participants) | 4 | 3
  4 Month : Ventilator | 0 | 1
  4 Month : Transfusion: number analyzed (Participants) | 4 | 3
  4 Month : Transfusion | 0 | 1
  4 Month : Antibiotics: number analyzed (Participants) | 4 | 3
  4 Month : Antibiotics | 1 | 1
  5 Month : Hospitalization: number analyzed (Participants) | 3 | 2
  5 Month : Hospitalization | 0 | 2
  5 Month : Ventilator: number analyzed (Participants) | 3 | 2
  5 Month : Ventilator | 0 | 0
  5 Month : Transfusion: number analyzed (Participants) | 3 | 2
  5 Month : Transfusion | 0 | 0
  5 Month : Antibiotics: number analyzed (Participants) | 3 | 2
  5 Month : Antibiotics | 0 | 1
  6 Month : Hospitalization: number analyzed (Participants) | 4 | 2
  6 Month : Hospitalization | 3 | 0
  6 Month : Ventilator: number analyzed (Participants) | 4 | 2
  6 Month : Ventilator | 0 | 0
  6 Month : Transfusion: number analyzed (Participants) | 4 | 2
  6 Month : Transfusion | 0 | 0
  6 Month : Antibiotics: number analyzed (Participants) | 4 | 2
  6 Month : Antibiotics | 1 | 0

3. Secondary Outcome: Cumulative Incidence of Documented Bacterial, Fungal, and Viral Infections
Description: Records will be assessed at baseline and prospectively while on study.
Time Frame: Baseline, up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I | Correlative
Number analyzed (Participants) | 4 | 5
Participants | 2 | 5

ADVERSE EVENTS:
Time Frame: 6 months
Description: only patients on Arm I (recieving drug on protocol) were tracked for toxicities
Arm/Group | Arm I | Control Arm | Correlative
Serious Adverse Events (participants affected / at risk) | 4/4 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 4/4 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (N=4) | Control Arm (N=0) | Correlative (N=0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (3) | 0 (0) | 0 (0)
hyperglycemia (Investigations) | 2 (6) | 0 (0) | 0 (0)
hyponatremia (Investigations) | 1 (1) | 0 (0) | 0 (0)
hypokalemia (Investigations) | 1 (1) | 0 (0) | 0 (0)
serum glutamic pyruvic transaminase (Investigations) | 1 (1) | 0 (0) | 0 (0)
Thrombosis/thrombus/embolism (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Heartburn/dyspepsia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Confusion (General disorders) | 1 (1) | 0 (0) | 0 (0)
"Distension bloating, abdominal" (General disorders) | 1 (1) | 0 (0) | 0 (0)
Infection Bladder (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lipase (Investigations) | 1 (1) | 0 (0) | 0 (0)
Lymphopenia (Investigations) | 1 (2) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infection Sinus (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils: Nose (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (N=4) | Control Arm (N=0) | Correlative (N=0)
Low WBC (Investigations) | 1 (1) | 0 (0) | 0 (0)
low Platelets (Investigations) | 3 (9) | 0 (0) | 0 (0)
Low Hemoglobin (Investigations) | 4 (15) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (3) | 0 (0) | 0 (0)
Anorexia (General disorders) | 2 (2) | 0 (0) | 0 (0)
Gastrointestinal - Other (General disorders) | 1 (1) | 0 (0) | 0 (0)
Alkaline phosphatase (Investigations) | 3 (10) | 0 (0) | 0 (0)
Creatinine (Investigations) | 2 (7) | 0 (0) | 0 (0)
Proteinuria (Investigations) | 2 (2) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Taste alteration (General disorders) | 1 (5) | 0 (0) | 0 (0)
Insomnia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Dermatology/Skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (2) | 0 (0) | 0 (0)
Weight loss (General disorders) | 1 (1) | 0 (0) | 0 (0)
hyperglycemia (Investigations) | 4 (15) | 0 (0) | 0 (0)
hypoglycemia (Investigations) | 1 (1) | 0 (0) | 0 (0)
hypocalcemia (Investigations) | 4 (4) | 0 (0) | 0 (0)
hypomagnesemia (Investigations) | 3 (3) | 0 (0) | 0 (0)
hyponatremia (Investigations) | 3 (7) | 0 (0) | 0 (0)
hypokalemia (Investigations) | 1 (3) | 0 (0) | 0 (0)
hypoalbuminemia (Investigations) | 4 (6) | 0 (0) | 0 (0)
hyperbilirubinemia (Investigations) | 1 (1) | 0 (0) | 0 (0)
serum glutamic pyruvic transaminase (Investigations) | 2 (10) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (4) | 0 (0) | 0 (0)
Pain: Head/headache (General disorders) | 1 (1) | 0 (0) | 0 (0)
serum glutamic oxaloacetic transaminase (Investigations) | 1 (6) | 0 (0) | 0 (0)
hypermagnesemia (Investigations) | 2 (4) | 0 (0) | 0 (0)
hyperkalemia (Investigations) | 1 (2) | 0 (0) | 0 (0)
Ocular/Visual - Other (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary frequency/urgency (General disorders) | 1 (1) | 0 (0) | 0 (0)
Renal/Genitourinary - Other (General disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 0 (0)
Intra-operative Injury (General disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal Soft Tissue - Other (General disorders) | 1 (1) | 0 (0) | 0 (0)
Dry mouth (General disorders) | 3 (3) | 0 (0) | 0 (0)
Dehydration (General disorders) | 2 (3) | 0 (0) | 0 (0)
Pruritus/itching (General disorders) | 1 (2) | 0 (0) | 0 (0)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 2 (5) | 0 (0) | 0 (0)
Pain: Abdomen (General disorders) | 1 (1) | 0 (0) | 0 (0)
Ataxia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Obstruction Bladder (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pain Bladder (General disorders) | 1 (1) | 0 (0) | 0 (0)
Amylase (Investigations) | 1 (2) | 0 (0) | 0 (0)
Bronchospasm wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Urine color change (General disorders) | 1 (1) | 0 (0) | 0 (0)
Dry eye syndrome (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Anal Incontinence (General disorders) | 1 (1) | 0 (0) | 0 (0)
gamma-Glutamyl transpeptidase (Investigations) | 1 (1) | 0 (0) | 0 (0)
Glomerular filtration rate (Investigations) | 2 (4) | 0 (0) | 0 (0)
Lipase (Investigations) | 1 (1) | 0 (0) | 0 (0)
Lymphopenia (Investigations) | 2 (4) | 0 (0) | 0 (0)
Memory impairment (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pain: Muscle (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pain Oral cavity (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pain: Extremity-limb (General disorders) | 1 (1) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 2 (3) | 0 (0) | 0 (0)
Allergic rhinitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperpigmentation (General disorders) | 1 (5) | 0 (0) | 0 (0)
Mucositis/stomatitis Oral cavity (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
blurred vision (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Hemorrhage GU: Urinary (Vascular disorders) | 1 (2) | 0 (0) | 0 (0)
Thrombosis/embolism (vascular access-related) (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Mucositis/stomatitis Oral cavity (Infections and infestations) | 3 (11) | 0 (0) | 0 (0)
Infection Lip perioral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Blood Infection with high grade neutropenia (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
adverse events were only tracked on Arm I

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes